CLINICAL TRIAL: NCT05666934
Title: Using Home-based Augmented Reality Storybook Training Modules for Facilitating Emotional Functioning and Socialization of Children With Autism Spectrum Disorder
Brief Title: Home-based Augmented Reality Storybook Training Modules for Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Ling-Yi Lin, Associate Professor, National Cheng Kung University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-107-066
Record Dates: First submitted 2022-12-18; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based Augmented Reality Storybook Training Module (Experimental): The children were entirely involved in this intervention program at home, with 20 minutes each time, 4 times a week for 8 weeks. The caregiver was required to perform the interactive picture book specified by the AR home training modules. During the process, the caregivers could directly contact the researcher by telephone and instant messaging for solving problems that occur during the interaction. The researcher and the caregiver consistently met once every two weeks. On the day of the meeting, the caregiver needs to prepare at least ten minutes of interactive video to discuss with the researcher. The researcher not only provides suggestions for caregiver interaction skills based on the video, in order to facilitate the child's interaction. The interaction strategies were also revised according to the interaction ability and special behavior problems of individual children.
  Interventions: Device: Augmented Reality Storybook

INTERVENTIONS:
Device: Augmented Reality Storybook — The AR system was developed using a Vuforia Engine Package for Unity (PTC Inc, San Diego, CA), which enabled to create an application for children to view a storybook in their own homes. The children and caregivers could view eight scenarios (receiving a praise, broken toys, waiting in line at the playground, getting a vaccination, waiting for watching a video, hitting someone in an accident, grabbing a toy, understanding another person's feelings) and learn strategies for emotional events reflected in the tablet (Figure 1). This AR application supports a tablet size of 10.4 inches and is equipped with a Samsung Galaxy Tab A7.

SUMMARY:
Autism spectrum disorder (ASD) is a lifelong neurodevelopmental disability with increasing prevalence worldwide. The main difficulties include poor social interaction and self-regulation skills. Effective interventions are required to improve the social interaction skills and emotional regulation of children with ASD. The present study involved developing and testing the feasibility and short-term efficacy of the home-based augmented reality (AR) training modules for preschool children with ASD. We recruited 15 children with ASD (3 to 5 years old). Wilcoxon signed rank test analysis was used to compare the differences in emotional functioning and adaptive behavior. Children received 8-week home-based AR training modules. Sessions were 20 minutes 4 times a week.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a lifelong neurodevelopmental disability with increasing prevalence worldwide. Its symptoms include limitations in social interaction and repetitive and restrictive behaviors. These symptoms may result in difficulties in participating in daily life and social activities across the lifespan. The main challenges include poor communication, social interaction, and emotional regulation skills that can limit and impair a person's everyday functioning. Many parents of children with ASD had an increased caregiver burden. In addition, the total lifetime cost of autism per individual is about 3.6 million US dollars. Thus, there is an urgent need to develop appropriate and effective interventions for improving the communication and self-regulation skills of children with ASD. Research has increasingly focused on the effectiveness of interventions for children with ASD. Nonetheless, research has yet remained an underappreciated concept in different cultural contexts. To address these gaps, the present study involved developing and testing the feasibility and effectiveness of the home-based Augmented Reality (AR) social story training modules for preschool children with ASD. The home-based AR social story training modules are designed. We recruited 15 children with ASD (3 to 5 years old). Wilcoxon signed rank test analysis was used to compare the differences in emotional functioning and adaptive behavior. Children received 8-week home-based AR training modules. Sessions were 20 minutes 4 times a week.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were children who (1) had a disability identification for ASD, (2) were aged 3 to 5 years and 11 months, and (3) scores at or above 30 according to the CARS-2.

Exclusion Criteria:

* The exclusion criteria were children (1) whose nonverbal intelligence quotient was below 85 and (2) who had comorbid diagnoses with attention deficit hyperactivity disorder (ADHD).

Ages: 41 Months to 70 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Vineland Adaptive Behavior Scales-Third Edition | 8 weeks
  The Vineland Adaptive Behavior Scales-Third Edition (VABS-3) comprises four domains, that is, communication, daily living skills, socialization and motor skills, for assessing adaptive functioning in children aged 3 to 12 years old. The raw score in each domain and total raw score are converted to an age-equivalent score. The domain scores are also expressed as standard scores with a mean of 100 and standard deviation of 15. The range for each subscale is from 20 to 140. The subscales are summed to compute a total score, ranging from 80 to 560. The higher the scores are, the better adaptive functioning the children achieve.
Functional Emotional Assessment Scale | 8 weeks
  The Functional Emotional Assessment Scale (FEAS; Greenspan et al., 2001) is based on six functional developmental levels of the developmental individual-difference relationship-based model and divided into two parts that (1) examine the children's development and (2) assess the parenting skills. All parents in the study were asked to record their parent-child activities as 15-minute videos. All videos were coded using random numbers to hide the research information (e.g. groups and test time). Two videos (pre- and post-test) were reviewed for each child. Using the Chinese version of the Scoring Form translated by Liao et al. (2014; intraclass correlation coefficient = 0.85), each item of the FEAS was rated as 0, 1 or 2. Higher raw scores represent better functions and skills. The total score is summed and ranges from 0 to 80.

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Yi Lin, ScD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No